CLINICAL TRIAL: NCT00051337
Title: The Physiology of Paroxysmal Hyperkinetic Movement Disorders: A SPECT Study
Brief Title: Single Photon Emission Computed Tomography (SPECT) to Study Paroxysmal Hyperkinetic Movement Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030072; 03-N-0072
Record Dates: First submitted 2003-01-08; First posted 2003-01-09 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Hyperkinesis
Keywords: Kinesiogenic; Psychogenic; Channelopathy; Ictal; Paroxysmal Dyskinesia; Psychogenic Movement Disorders; Single Photon Emission; Computed Tomography (SPECT)
MeSH Terms: conditions — Hyperkinesis; Channelopathies; Chorea

SUMMARY:
This study will use single photon emission computed tomography (SPECT) to determine what areas of the brain are responsible for paroxysmal hyperkinetic movement disorders. Patients with these disorders have sudden, brief attacks of movement, similar to epileptic seizures, but without loss of consciousness. SPECT is a nuclear medicine test that produces three-dimensional images of the brain, showing blood flow and function in different brain regions. This test, which can detect the focus of epileptic seizures, will be used in this study to scan patients while they are experiencing a hyperkinetic movement attack, while they are not having and attack, and while they are simulating an attack.

Patients 18 years of age and older who have paroxysmal movement attacks that can be easily induced by a specific trigger, such as a sudden movement or prolonged exercise, may be eligible for this study. Candidates will be screened with a medical history and review of their medical records, physical examination, videotape of attacks, and, for women, a pregnancy test.

Participants will have three SPECT scans, separated from each other by at least 48 hours. Before each scan, the subject will perform an activity that ordinarily precipitates a movement attack, such as standing up from a chair, assuming a certain posture, or doing something strenuous. Each scan will try to record one of the following conditions:

* The subject performs the trigger activity, but does not have an attack;
* The subject performs the trigger activity and has an involuntary attack as a result;
* The subject performs the trigger activity and does not have an attack, but then mimics an attack voluntarily.

After the condition is recorded, the subject will be given an injection of a radioactive agent called 99m Technetium and will then relax quietly for 40 to 60 minutes before the SPECT scan. For the scan, the subject lies on an examination table and the SPECT camera is moved near and around the head to image the brain. The scan takes about 40 minutes.

Participants will also undergo one magnetic resonance imaging (MRI) scan. For this test, the subject lies in a narrow cylinder (the scanner), while pictures of the brain are taken. Earplugs are worn to muffle loud noises caused by electrical switching of radio frequency circuits used in the scanning process. The procedure takes about 30 minutes.

DETAILED DESCRIPTION:
The purpose of this study is to determine the areas of the brain responsible for paroxysmal hyperkinetic movement disorders. Paroxysmal hyperkinetic movement disorders have been clinically recognized for a long time, although the exact neurophysiological mechanism leading to paroxysms of hyperkinetic movement attacks is not well understood. Paroxysmal hyperkinetic movement disorders are heterogenous, and the exact mechanism may differ in each subcategory. In paroxysmal dyskinesias, the idiopathic forms of paroxysmal hyperkinetic movement disorders, it is speculated that transient functional abnormality at the cellular level occurs in the basal ganglia without organic irreversible damage. Ion channel dysfunction is an attractive hypothesis to explain such transient dysfunction. Some patients with paroxysmal hyperkinetic movement disorders have a psychogenic etiology.

A promising technique to evaluate physiological changes in the brain during an attack is ictal single photon emission computed tomography (SPECT) scanning. Ictal SPECT is a reliable method to detect a seizure focus during an epileptic seizure. We will utilize ictal SPECT scanning techniques during, and between attacks, and while they are simulating such attacks. The differential activation between the attacks of hyperkinetic movements and the voluntary movements may shed light on the regions of the brain and neurophysiological mechanisms responsible for generation of paroxysmal hyperkinetic movement disorders.

ELIGIBILITY:
INCLUSION CRITERIA - Paroxysmal Dyskinesia Patients:

Established diagnosis of paroxysmal hyperkinetic movement disorders. The diagnosis will be established by the preliminary screening in the NINDS Movement Disorders Outpatient Clinic, based on review of medical record, history, clinical evaluation, and video tapes of an attack.

Age 18 or older.

A reproducible trigger of paroxysmal hyperkinetic attacks, such as sudden movement, or prolonged exercise, which will produce attacks at least with 50% consistency.

Patients only with paroxysmal attacks of hyperkinetic movements.

Patients whose attacks can be precipitated easily.

Patients whose typical attack last at least 15 seconds.

Patients taking medication that may influence the central nervous system, such as phenytoin, phenobarbital, carbamazepine, clonazepam, and antidepressants (but not limited to these) for their paroxysmal dyskinesias (not seizures) will be asked to hold the medication prior to the study. A sufficient drug washout period will be established dependant upon the individual drug. Subjects may be admitted to the NIH if necessary. They will be asked to abstain from alcohol and caffeine 24 hours prior to the study as well.

INCLUSION CRITERIA - Psychogenic paroxysmal hyperkenetic movement attack patients:

Established diagnosis of psychogenic hyperkinetic movement disorders. The diagnosis will be established by the preliminary screening in the NINDS Movement Disorders Outpatient Clinic, based on review of medical record, history, clinical evaluation, and video tapes of an attack.

Patients with clear onset, stereotyped, defined and evaluable hyperkinetic attacks.

Patients only with paroxysmal attacks of hyperkinetic movements.

Age 18 or older.

A reproducible trigger of paroxysmal hyperkinetic attacks, such as sudden movement, startle or prolonged exercise, which will produce attacks at least with 50% consistency.

Patients whose attacks can be precipitated easily.

Patients whose typical attack last at least 15 seconds.

Patients taking medication that may influence the central nervous system, such as phenytoin, phenobarbital, carbamazepine, clonazepam, and antidepressants (but not limited to these) will be asked to hold the medication prior to the study. A sufficient drug washout period will be established dependant upon the individual drug. Subjects may be admitted to the NIH if necessary. They will be asked to abstain from alcohol and caffeine 24 hours prior to the study as well.

EXCLUSION CRITERIA:

Age younger than 18 years old.

Previous history of or MRI findings consistent with brain tumors, strokes, trauma or arterial venous malformations.

Contraindication to MRI such as having devices not compatible with MRI (pacemaker, an implanted medical pump, brain stimulators etc.), metallic prostheses in their body (metal pins and rods, heart valves, cochlear implants etc.), and history of working with metals in the past, since such persons may potentially have small metal fragments in the eye without being aware of it.

Any diagnosis of progressive neurological disorders other than paroxysmal hyperkinetic movement disorder.

Any history of significant medical disorders requiring chronic treatment with other drugs that affect the CNS, which cannot be stopped.

Ongoing radiation therapy for medical condition such as cancer.

Women who are pregnant or nursing. Female subjects of child bearing potential will have specific interview and a pregnancy test prior to the study (before each imaging procedure if required) to ensure that they are not pregnant or nursing.

Any subject who is not capable of giving an informed consent. This will be determined at the initial evaluation at NINDS clinic. Patients with Mini Mental Score less than 25 or significant psychiatric history will be further evaluated by detailed neuropsychiatric testing, or consultation with a psychiatrist.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Demirkiran M, Jankovic J. Paroxysmal dyskinesias: clinical features and classification. Ann Neurol. 1995 Oct;38(4):571-9. doi: 10.1002/ana.410380405. PMID 7574453
- [Background] Kertesz A. Paroxysmal kinesigenic choreoathetosis. An entity within the paroxysmal choreoathetosis syndrome. Description of 10 cases, including 1 autopsied. Neurology. 1967 Jul;17(7):680-90. doi: 10.1212/wnl.17.7.680. No abstract available. PMID 6067487
- [Background] Stevens H. Paroxysmal choreo-athetosis. A form of reflex epilepsy. Arch Neurol. 1966 Apr;14(4):415-20. doi: 10.1001/archneur.1966.00470100071009. No abstract available. PMID 5906466